CLINICAL TRIAL: NCT07127692
Title: Exploratory Study on the Prevalence of Sarcopenia-Promoting Medicines in Patients With Sarcopenia and Falls
Brief Title: Prevalence of Sarcopenia-Promoting Medicines in Patients With Sarcopenia and Falls
Status: Not yet recruiting | Type: Observational
Sponsor: Medway NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Kamaldeep Sahota, Lead Clinical Pharmacist Frailty, Medway NHS Foundation Trust
Other Study IDs: 354863
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia in Elderly; Falls
Keywords: Sarcopenia-promoting medicines; Sarcopenia; Falls; Medicines in elderly
MeSH Terms: conditions — Sarcopenia | interventions — Insemination, Artificial, Heterologous; Walking; Hand Strength; Walking Speed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Strength, Assistance with walking, Rise from a chair, Climb stairs, and Falls (SARC-F) questionnaire — Self-administered screening tool for sarcopenia
Diagnostic Test: Hand grip strength — Used to assess sarcopenia
Diagnostic Test: Timed Up and Go test — Screening test for falls in elderly
Diagnostic Test: Gait speed — Assessment to check for functional mobility and risk of falls.
Diagnostic Test: Clinical Frailty Scale (CFS) — Used to assess level of frailty.

SUMMARY:
Sarcopenia, characterised by the loss of muscle mass and function, is a common condition among the elderly and is often associated with increased risk of falls. Certain medications, such as glucocorticoids, statins, and some antipsychotics, may exacerbate sarcopenia, leading to a higher incidence of falls. This study aims to explore the prevalence of such medicines in patients diagnosed with sarcopenia who have experienced falls. Understanding the impact of these medications on sarcopenia and fall risk can inform clinical guidelines and improve patient outcomes.

DETAILED DESCRIPTION:
Sarcopenia, the age-related loss of muscle mass and strength, is a recognised contributor to frailty, disability, and increased fall risk in older adults. While physical inactivity and comorbidities are known risk factors, increasing evidence suggests that certain medications - including corticosteroids, sedatives and statins - may also contribute to muscle decline. These medicines are frequently prescribed to older adults, but the extent of their use in patients with sarcopenia and falls remains poorly defined.

Falls clinics manage high-risk patients, yet there is currently limited research examining the prevalence of sarcopenia-promoting medications in this specific setting. This study addresses an important knowledge gap by estimating the prevalence of these medicines in older adults attending a secondary care falls clinic, and by exploring associations with sarcopenia and fall history.

The findings will support a better understanding of medication-related risk factors for sarcopenia and may help guide future deprescribing and medication review strategies. This aligns with current priorities in geriatric medicine to reduce inappropriate polypharmacy and improve outcomes for older adults through targeted, evidence-based prescribing.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥65 years
* Attendance at the falls clinic for a new assessment
* Diagnosed with sarcopenia (based on the European Working Group on Sarcopenia in Older People (EWGSOP2) criteria)
* History of falls in the past 12 months

Exclusion Criteria:

* Cognitive impairment preventing consent
* Acute medical instability
* Enrolled in on other clinical trials.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will be conducted in a multidisciplinary falls clinic at Medway NHS Foundation Trust, based in Gillingham, Kent, England, UK. This secondary care setting receives referrals primarily from inpatient hospital teams and primary care practitioners. The clinic routinely assesses older adults who have experienced falls or are at high risk of falling, and conducts comprehensive geriatric assessments, including medication reviews, functional status evaluations, and frailty assessments.
Sampling Method: Non-Probability Sample
Enrollment: 323 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of exposure to one or more sarcopenia-promoting medication | 6 months
  Proportion of adults aged 65 years and over attending the falls clinic who are prescribed one or more sarcopenia-promoting medication. Unit of measure: % of participants.

SECONDARY OUTCOMES:
Distribution of sarcopenia-promoting medication classes | 6 months
  Proportion of participants exposed to each medication class. Unit of measure: % of participants per medication class.
Number of sarcopenia-promoting medications per participant | 6 months
  Mean number of eligible medications prescribed per participant. Unit of measure: count.
Handgrip strength | 6 months
  Mean maximum grip strength measured with a Jamar dynamometer. Unit of Measure: Kilograms (kg).
Gait speed | 6 months
  Mean walking speed measured over 4 metres. Unit of measure: metres per second (m/s)
SARC-F score | 6 months
  SARC-F mean score. Unit of measure: points (0-10)
Timed Up and Go Test | 6 months
  Mean time taken to stand from a chair, walk 3 metres, turn, walk back and sit down. Unit of measure: Seconds (s).
Association between medication burden and functional performance | 6 months
  Comparison of grip strength, gait speed, SARC-F scores and Timed Up and Go performance across groups defined by medication burden e.g. 0-1 vs >2 sarcopenia promoting medications. Units of measure: Differences in mean values (kg, m/s, points, seconds).

CONTACTS AND LOCATIONS:
Overall Officials: Kamaldeep K Sahota, Pharmacist, Principal Investigator — Medway NHS Foundation Trust
Locations (1):
- Medway NHS Foundation Trust, Gillingham, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zia A, Kamaruzzaman SB, Tan MP. Polypharmacy and falls in older people: Balancing evidence-based medicine against falls risk. Postgrad Med. 2015 Apr;127(3):330-7. doi: 10.1080/00325481.2014.996112. Epub 2014 Dec 24. PMID 25539567
- [Result] Veronese, N., et al. (2020). Polypharmacy is associated with higher frailty risk in older people: A systematic review and meta-analysis. Journal of the American Medical Directors Association, 21(2), 181-187.
- [Result] Tanskanen, A., et al. (2015). Anticholinergic burden and physical functioning in older people: A systematic review. Drugs & Aging, 32(10), 741-750.
- [Result] Shafiee G, Keshtkar A, Soltani A, Ahadi Z, Larijani B, Heshmat R. Prevalence of sarcopenia in the world: a systematic review and meta- analysis of general population studies. J Diabetes Metab Disord. 2017 May 16;16:21. doi: 10.1186/s40200-017-0302-x. eCollection 2017. PMID 28523252
- [Result] Scott, D., et al. (2016). Sarcopenia and statin use: A potential link? Drugs & Aging, 33(1), 1-9.
- [Result] Reeve E, Wiese MD, Hendrix I, et al. (2014). The impact of deprescribing interventions on polypharmacy and clinical outcomes: a systematic review and meta-analysis. J Am Med Dir Assoc. 15(3):131-6. https://doi.org/10.1016/j.jamda.2013.11.008
- [Result] Rawle MJ, Westbury LD, Russell S, et al (2018). Anticholinergic drug burden and cognitive function in people aged 50 years and older: the English Longitudinal Study of Ageing. Age Ageing; 47(4):505-11 https://doi.org/10.1093/ageing/afy026
- [Result] Perlman C, Kirkham J, Velkers C, Leung RH, Whitehead M, Seitz D. Access to Psychiatrist Services for Older Adults in Long-Term Care: A Population-Based Study. J Am Med Dir Assoc. 2019 May;20(5):610-616.e2. doi: 10.1016/j.jamda.2019.01.121. Epub 2019 Mar 1. PMID 30827894
- [Result] Landi F, Liperoti R, Russo A, Giovannini S, Tosato M, Capoluongo E, Bernabei R, Onder G. Sarcopenia as a risk factor for falls in elderly individuals: results from the ilSIRENTE study. Clin Nutr. 2012 Oct;31(5):652-8. doi: 10.1016/j.clnu.2012.02.007. Epub 2012 Mar 11. PMID 22414775
- [Result] Fox C, Richardson K, Maidment ID, Savva GM, Matthews FE, Smithard D, Coulton S, Katona C, Boustani MA, Brayne C. Anticholinergic medication use and cognitive impairment in the older population: the medical research council cognitive function and ageing study. J Am Geriatr Soc. 2011 Aug;59(8):1477-83. doi: 10.1111/j.1532-5415.2011.03491.x. Epub 2011 Jun 24. PMID 21707557
- [Result] Cruz-Jentoft AJ, Bahat G, Bauer J, Boirie Y, Bruyere O, Cederholm T, Cooper C, Landi F, Rolland Y, Sayer AA, Schneider SM, Sieber CC, Topinkova E, Vandewoude M, Visser M, Zamboni M; Writing Group for the European Working Group on Sarcopenia in Older People 2 (EWGSOP2), and the Extended Group for EWGSOP2. Sarcopenia: revised European consensus on definition and diagnosis. Age Ageing. 2019 Jul 1;48(4):601. doi: 10.1093/ageing/afz046. No abstract available. PMID 31081853
- [Result] Corsonello A, Pedone C, Incalzi RA. Age-related pharmacokinetic and pharmacodynamic changes and related risk of adverse drug reactions. Curr Med Chem. 2010;17(6):571-84. doi: 10.2174/092986710790416326. PMID 20015034

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT07127692/Prot_SAP_000.pdf
  • Informed Consent Form (2025-07-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT07127692/ICF_001.pdf